CLINICAL TRIAL: NCT00430404
Title: Randomized Controlled Trial of a Community-based Early Psychiatric Intervention Strategy to Screen and Manage Depression in the Elderly
Brief Title: Screening and Treatment of Depression in the Community
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: National University Hospital, Singapore (Other)
Collaborators: National University of Singapore (Other)
Responsible Party: Principal Investigator, Psychological Medicine, Ng Tz Pin, MD, MFPHM, National University Hospital, Singapore, National University Hospital, Singapore
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: NMRC/0846/2004
Record Dates: First submitted 2007-01-31; First posted 2007-02-01 (Estimated); Last update posted 2014-01-03 (Estimated); Status verified 2014-01

CONDITIONS: Depression
MeSH Terms: conditions — Depression | interventions — Methods

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Usual care (controlled group) (No Intervention): Usual care for management of depression
- collaborative care (Intervention) (Experimental): Collaborative care for management of depression for intervention group. We provided multidisciplinary groups of care from psychiatrist, psychologist, social counselor, general practitioners and case managers for intervention group.
  Interventions: Other: Collaborative care (Intervention)

INTERVENTIONS:
Other: Collaborative care (Intervention) — Structured shared care with treatment protocol & support
  Other Names: Community based early psychiatric intervention strategy
  Arms: collaborative care (Intervention)

SUMMARY:
To evaluate the effectiveness of a community-based strategy of routine population mass screening for depression with follow-up feedback and management in a primary care non-psychiatric setting involving a structured, multifaceted, collaborative (primary care and hospital-based)shared care programme.

Hypotheses:

We hypothesize that a community-based early psychiatric interventional strategy (CEPIS) for depression in the elderly leads to increased recognition of depression by primary care physicians, more initiation of treatment for emotional problems, and improved outcomes for patients with depression, as measured by:

1. increased rates of detection or recognition by a primary care physician of minor or major (clinical) depression.
2. higher rates of management activities: counselling for psychological, family social problems, contact with community family services (human service agency), consultation and/or referral to a mental health specialist
3. Reduced depressive symptom severity, improved level of daily functioning and quality of life among those with major clinical depression
4. Better patient satisfaction with care
5. Favourable clinician's and patients perception of their usefulness or acceptability

DETAILED DESCRIPTION:
Depression is a highly prevalent, clinically under-recognized and under-treated medical disorder world wide. In Singapore, 17% of the adult population experience recent psychiatric disturbances, yet only 6% use the services of any health professional. General practitioners are the most commonly preferred caregiver, and actually used by 41.1% of those who sought help. At the same time, suicide rates especially among the elderly remain at very high levels compared to other countries in the world.

In recent decades, screening questionnaires have been developed and validated that are suitable for the initial detection of depression in the primary care setting. Previous research have shown that screening for depression do not result in increased recognition rates of mental disorders unless positive cases are selectively fed back to primary care physicians. They also do not translate into increased rates of interventional activities such as initiation of therapy and referral to mental health specialists. Neither dose primary care physician education or clinical practice guidelines result in any improved outcomes for the patients unless these are accompanied by more sophisticated strategies in the organization and delivery of care, such as structured, collaborative, multidisciplinary care together with quality improvement processes.

More empirical data are therefore needed to establish whether screening for psychiatric disorders will enhance the recognition of clinical disorder, leading to better patient outcomes.

ELIGIBILITY:
Inclusion Criteria:

* > 60 years without dementia,
* Major depressive disorder,
* Bipolar disorder,
* Dysthymia disorder,
* Anxiety disorder,
* Mania/hypomania

Exclusion Criteria:

* Severe post-stroke dementia or aphasia,
* History of mania, psychiatric consultation or admission to hospital in past 3 months,
* MMSE score <18,
* Fully dependent at 3 or more basic activities of daily living,
* Very high BDI score (>=30),
* Serious suicidal risk,
* Current psychotic symptoms,
* Current alcohol abuse,
* Very high GDS score (>=12) confirmed by SCID

Min Age: 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 214 (Actual)
Dates: Start 2004-08; Primary Completion 2007-08 (Actual); Study Completion 2007-09 (Actual)

PRIMARY OUTCOMES:
Response to treatment at 6 months follow up is defined as a 50% reduction in HAMD-17 score | 6 months
  After enrolled in the study for 6 months, depressive symptoms were expected to reduce to 50% in assessment fo HAM_D 17

SECONDARY OUTCOMES:
Rates of physician and patient self-report of service utilization at 6 month follow up | 6 months
  Report of primary care physicians and patient's self report of using of health service for the treatment of depression
Improvement in follow-up SF-12 scores from baseline | 12 months
  Study participants' physical component and mental component of Quality of life were assessed after 12 months.
Caregiver burden at 6 month follow-up | 6 months
  Caregiver burden on taking care of depressive patients was assessed after 6months of study.
Patient satisfaction with care at 6 month follow up | 6 months
  Participants under intervention care (collaborative care) were surveyed about their satisfaction with the program after 6 months of enrollment in the study.
Physician feedback at 6 month follow up | 6 months
  primary physicians in the both arms were surveyed for their satisfaction about the study programme after the 6 months of study.

CONTACTS AND LOCATIONS:
Overall Officials: Ng Tz Pin, MD,MFPHM, Principal Investigator — Gerontological Research Programme, Faculty of Medicine, National University of Singapore
Locations (1):
- Department of Psychological Medicine, National University Hospital, 5 Lower Kent Ridge Road, Singapore, Singapore